CLINICAL TRIAL: NCT03745638
Title: A Phase 3, Double-Blind, Randomized, 8-Week, Vehicle-Controlled Efficacy and Safety Study of Ruxolitinib Cream Followed by a Long-Term Safety Extension Period in Adolescents and Adults With Atopic Dermatitis
Brief Title: Topical Ruxolitinib Evaluation in Atopic Dermatitis Study 1 (TRuE AD1) - An Efficacy and Safety Study of Ruxolitinib Cream in Adolescents and Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 18424-303; 2018-003712-45 (EudraCT Number)
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Pruritus; Eczema; Topical Therapy; JAK Inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- VC Period: Vehicle Cream BID (Placebo Comparator): Participants received vehicle cream, applied topically to the affected areas as a thin film twice daily (BID) from Day 1 to Week 8 during the Vehicle Control (VC) Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
  Interventions: Drug: Vehicle Cream
- VC Period: Ruxolitinib 0.75% Cream BID (Experimental): Participants received ruxolitinib 0.75% cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 8 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
  Interventions: Drug: Ruxolitinib Cream
- VC Period: Ruxolitinib 1.5% Cream BID (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 8 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
  Interventions: Drug: Ruxolitinib Cream
- LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID (Experimental): Participants who applied vehicle cream BID during the VC Period, were randomized to apply ruxolitinib 0.75% cream, topically to the affected areas as a thin film BID from Week 8 to 52 during the Long-term Safety (LTS) Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
  Interventions: Drug: Ruxolitinib Cream
- LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID (Experimental): Participants who applied vehicle cream BID during the VC Period, were randomized to apply ruxolitinib 1.5% cream, topically to the affected areas as a thin film BID from Week 8 to 52 during the LTS Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
  Interventions: Drug: Ruxolitinib Cream
- LTS Period: Ruxolitinib 0.75% Cream (Experimental): Arm description: Participants who applied ruxolitinib 0.75% cream during VC Period, continued applying ruxolitinib 0.75% cream topically to the affected areas as a thin film BID from Week 8 to 52 during the LTS Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
  Interventions: Drug: Ruxolitinib Cream
- LTS Period: Ruxolitinib 1.5% Cream (Experimental): Arm description: Participants who applied ruxolitinib 1.5% cream during VC Period, continued applying ruxolitinib 1.5% cream topically to the affected areas as a thin film BID from Week 8 to 52 during the LTS Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
  Interventions: Drug: Ruxolitinib Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream applied topically to the affected area as a thin film twice daily.
  Other Names: INCB018424 Phosphate Cream
  Arms: LTS Period: Ruxolitinib 0.75% Cream; LTS Period: Ruxolitinib 1.5% Cream; LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID; LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID; VC Period: Ruxolitinib 0.75% Cream BID; VC Period: Ruxolitinib 1.5% Cream BID
Drug: Vehicle Cream — Matching vehicle cream applied topically to the affected area as a thin film twice daily.
  Arms: VC Period: Vehicle Cream BID

SUMMARY:
The purpose of this study is to assess the efficacy and safety of twice daily ruxolitinib cream in adolescents and adults with Atopic Dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged ≥12 to 17 years, inclusive, and men and women aged ≥18 years.
* Participants diagnosed with Atopic Dermatitis (AD) as defined by the Hanifin and Rajka criteria.
* AD duration of at least 2 years.
* Participants with an Investigator's Global Assessment (IGA) score of 2 to 3 at screening and Baseline [Vehicle Controlled (VC) Period] and 0 to 4 at Week 8 [Long-Term Safety (LTS) Period].
* Participants with percentage of Body Surface Area (% BSA) (excluding scalp) of AD involvement of 3% to 20% at screening and Baseline (VC Period) and 0% to 20% at Week 8 (LTS Period).
* Participants who agree to discontinue all agents used to treat AD from screening through the final follow-up visit.
* Participants who have at least 1 "target lesion" that measures approximately 10 cm^2 or more at screening and Baseline. Lesion must be representative of the participant's disease state and not be located on the hands, feet, or genitalia.
* Willingness to avoid pregnancy or fathering of children.

Exclusion Criteria:

* Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to Baseline.
* Concurrent conditions and history of other diseases:

  * Immunocompromised.
  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before Baseline.
  * Active acute bacterial, fungal, or viral skin infection within 1 week before Baseline.
  * Any other concomitant skin disorder, pigmentation, or extensive scarring that, in the opinion of the investigator, may interfere with the evaluation of AD lesions or compromise participant safety.
  * Presence of AD lesions only on the hands or feet without prior history of involvement of other classical areas of involvement such as the face or the folds.
  * Other types of eczema.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Use of any of the following treatments within the indicated washout period before Baseline:

  * 5 half-lives or 12 weeks, whichever is longer - biologic agents (eg. dupilumab).
  * 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs, cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg. mycophenolate or tacrolimus).
  * 2 weeks - immunizations and sedating antihistamines, unless on long-term stable regimen (nonsedating antihistamines are permitted).
  * 1 week - use of other topical treatments for AD (other than bland emollients). Diluted sodium hypochlorite "bleach" baths are allowed as long as they do not exceed 2 baths per week and their frequency remains the same throughout the study.
* Participants who have previously received Janus kinase (JAK) inhibitors, systemic or topical.
* Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation within 2 weeks prior to Baseline and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the participant's AD.
* Positive serology test results at screening for Human Immunodeficiency Virus (HIV) antibody.
* Liver function tests: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 × upper limit of normal (ULN); alkaline phosphatase and/or bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Pregnant or lactating participants, or those considering pregnancy.
* History of alcoholism or drug addiction within 1 year before screening or current alcohol or drug use that, in the opinion of the investigator, will interfere with the participant's ability to comply with the administration schedule and study assessments.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before Baseline with another investigational medication or current enrollment in another investigational drug protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Kuligowski, MD, PhD, MBA, Study Director — Incyte Corporation
Locations (79):
- United States (42):
  - Cahaba Dermatology, Birmingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists Inc, Oceanside, California
  - Integrated Research Group Inc., Riverside, California
  - Advanced Rx Clinical Research, Westminster, California
  - Clearlyderm Boca Raton - BTC - PPDS, Boca Raton, Florida
  - Olympian Clinical Research, Largo, Florida
  - Acevedo Clinical Research, Miami, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - AdvancedPharma CR LLC, Miami, Florida
  - University of South Florida, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Aeroallergy Research Lab Of Savannah, Savannah, Georgia
  - Clinical Research Atlanta - ERN-PPDS, Stockbridge, Georgia
  - Sneeze Wheeze and Itch Associates LLC, Normal, Illinois
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - DS Research, New Albany, Indiana
  - Kansas City Dermatology P.A., Overland Park, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Michael W Simon MD, Nicholasville, Kentucky
  - DermAssociates, Rockville, Maryland
  - Henry Ford Medical Center, Detroit, Michigan
  - JDR Dermatology Research, Las Vegas, Nevada
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Sadick Dermatology, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Ohio Pediatric Research Assn Inc, Huber Heights, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Cyn3rgy Research - Clinedge - PPDS, Gresham, Oregon
  - Clinical Research Institute Of Southern Oregon - Crisor, Medford, Oregon
  - Oregon Medical Research Center PC, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Synexus Clinical Research Us Inc. Greer, Greer, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Family Medicine Associates Of Texas, Carrollton, Texas
  - Progressive Clinical Research PA, San Antonio, Texas
  - Jordan Valley Medical Center, West Jordan, Utah
  - PI Coor Clinical Research LLC, Burke, Virginia
  - West End Dermatology, Henrico, Virginia
- Canada (6):
  - Lynderm Research Inc, Markham, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Siena Medical Reserch Corporation, Westmount, Quebec
- France (5):
  - CHRU de Brest - Hopital Morvan, Brest
  - Le Bateau Blanc - Imm. A, Martigues
  - Hôpital L'archet 2, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Charles Nicolle, Rouen
- Germany (5):
  - Elben Klinken Stade - Buxtehude, Buxtehude, Lower Saxony
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Universitatsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Frankfurt, Frankfurt am Main
- Hungary (6):
  - Synexus (DRS) - Synexus Magyarország Kft. Budapest, Budapest
  - Synexus Affiliate - Synexus Magyarorszag Kft. Debrecen, Debrecen
  - Synexus (DRS) - Synexus Magyarország Kft. Gyula, Gyula
  - Pécsi Tudományegyetem, Pécs
  - Allergo-Derm Bakos Kft., Szolnok
  - Synexus (DRS) - Synexus Magyarország Kft. Zalaegerszeg, Zalaegerszeg
- Fondazione Policlinico Universitario A Gemelli, Roma, Italy
- Poland (14):
  - Synexus - Wroclaw, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne ADAMAR, Wroclaw, Lower Silesian Voivodeship
  - ETG Zgierz, Zgierz, Lódzkie
  - Klinika Ambroziak, Warsaw, Masovian Voivodeship
  - Synexus - Gdansk, Gdansk, Pomeranian Voivodeship
  - Laser Clinic S.C., Szczecin, West Pomeranian Voivodeship
  - Synexus - Katowice, Katowice
  - Centrum Medyczne Krakow - PRATIA - PPDS, Krakow
  - ETG Lublin, Lublin
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z.o.o, Tarnów
  - Medycyna Kliniczna Marzena Waszczak-Jeka, Warsaw
  - ETG Warszawa, Warsaw
  - Royalderm, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simpson EL, Augustin M, Thaci D, Misery L, Armstrong AW, Blauvelt A, Papp KA, Szepietowski JC, Boguniewicz M, Kwatra SG, Kallender H, Sturm D, Ren H, Kircik L. Ruxolitinib Cream Monotherapy Improved Symptoms and Quality of Life in Adults and Adolescents with Mild-to-Moderate Atopic Dermatitis: Patient-Reported Outcomes from Two Phase III Studies. Am J Clin Dermatol. 2025 Jan;26(1):121-137. doi: 10.1007/s40257-024-00901-z. Epub 2024 Nov 15. PMID 39546129
- [Derived] Blauvelt A, Kallender H, Sturm D, Li Q, Ren H, Eichenfield LF. Efficacy and Safety of Ruxolitinib Cream in Atopic Dermatitis Based on Previous Medication History. Dermatol Ther (Heidelb). 2024 Nov;14(11):3161-3174. doi: 10.1007/s13555-024-01272-3. Epub 2024 Oct 7. PMID 39375281
- [Derived] Eichenfield LF, Simpson EL, Papp K, Szepietowski JC, Blauvelt A, Kircik L, Silverberg JI, Siegfried EC, Kuligowski ME, Venturanza ME, Kallender H, Ren H, Paller AS. Efficacy, Safety, and Long-Term Disease Control of Ruxolitinib Cream Among Adolescents with Atopic Dermatitis: Pooled Results from Two Randomized Phase 3 Studies. Am J Clin Dermatol. 2024 Jul;25(4):669-683. doi: 10.1007/s40257-024-00855-2. Epub 2024 May 2. PMID 38698175
- [Derived] Bloudek L, Eichenfield LF, Silverberg JI, Joish VN, Lofland JH, Sun K, Augustin M, Migliaccio-Walle K, Sullivan SD. Impact of Ruxolitinib Cream on Work Productivity and Activity Impairment and Associated Indirect Costs in Patients with Atopic Dermatitis: Pooled Results From Two Phase III Studies. Am J Clin Dermatol. 2023 Jan;24(1):109-117. doi: 10.1007/s40257-022-00734-8. Epub 2022 Oct 20. PMID 36264430
- [Derived] Gong X, Chen X, Kuligowski ME, Liu X, Liu X, Cimino E, McGee R, Yeleswaram S. Pharmacokinetics of Ruxolitinib in Patients with Atopic Dermatitis Treated With Ruxolitinib Cream: Data from Phase II and III Studies. Am J Clin Dermatol. 2021 Jul;22(4):555-566. doi: 10.1007/s40257-021-00610-x. Epub 2021 May 12. PMID 33982267
- [Derived] Papp K, Szepietowski JC, Kircik L, Toth D, Eichenfield LF, Leung DYM, Forman SB, Venturanza ME, Sun K, Kuligowski ME, Simpson EL. Efficacy and safety of ruxolitinib cream for the treatment of atopic dermatitis: Results from 2 phase 3, randomized, double-blind studies. J Am Acad Dermatol. 2021 Oct;85(4):863-872. doi: 10.1016/j.jaad.2021.04.085. Epub 2021 May 4. PMID 33957195
- [Derived] Scuron MD, Fay BL, Connell AJ, Peel MT, Smith PA. Ruxolitinib Cream Has Dual Efficacy on Pruritus and Inflammation in Experimental Dermatitis. Front Immunol. 2021 Feb 15;11:620098. doi: 10.3389/fimmu.2020.620098. eCollection 2020. PMID 33658996
- See also: Plain Language Summary of Results — http://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217471&parentIdentifier=INCB%2018424-303&attachmentIdentifier=2e6d9279-95cb-4501-9243-8a7bec8f8514&fileName=INCB18424-303_Plain_Language_Summary.pdf&versionIdentifier=6d478571-324e-42b3-b2cc-0d7125ac1386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 631 participants took part in the study at 78 sites, 48 in North America and 30 in Europe from December 20, 2018 to December 01, 2020.
Pre-assignment Details: Participants who completed Week 8 assessments of the Vehicle Control (VC) Period with no safety concerns continued in the 44-week Long Term Safety (LTS) Period. Participants who were on active treatment during the VC Period continued with the same treatment regimen in the LTS Period and those who applied vehicle cream during the VC Period were equally randomized into 1 of the 2 active treatment groups: ruxolitinib 0.75%, ruxolitinib 1.5% cream during the LTS Period.
Groups:
- VC Period: Vehicle Cream BID: Participants received vehicle cream, applied topically to the affected areas as a thin film twice daily (BID) from Day 1 to Week 8 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
- LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID: Participants who applied vehicle cream BID during the VC Period, were randomized to apply ruxolitinib 0.75% cream, topically to the affected areas as a thin film BID from Week 8 to 52 during the LTS Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Ruxolitinib 0.75% Cream: Participants who applied ruxolitinib 0.75% cream during VC Period, continued applying ruxolitinib 0.75% cream topically to the affected areas as a thin film BID from Week 8 to 52 during the LTS Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
- LTS Period: Ruxolitinib 1.5% Cream: Participants who applied ruxolitinib 1.5% cream during VC Period, continued applying ruxolitinib 1.5% cream topically to the affected areas as a thin film BID from Week 8 to 52 during the LTS Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
Period: Vehicle Control Period (Day 1 to Week 8)
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Started | 126 | 252 | 253 | 0 | 0 | 0 | 0
Completed | 95 | 222 | 225 | 0 | 0 | 0 | 0
Not Completed | 31 | 30 | 28 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 12 | 8 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 11 | 19 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 2 | 1 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Safety Period (Weeks 8 to 52)
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Started | 0 | 0 | 0 | 48 | 47 | 222 | 225
Completed | 0 | 0 | 0 | 37 | 38 | 176 | 174
Not Completed | 0 | 0 | 0 | 11 | 9 | 46 | 51
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 6 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 5 | 13 | 24
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 7 | 3 | 17 | 21
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized to the study.
Groups:
- VC Period: Vehicle Cream BID: Participants received vehicle cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 8 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
- Total: Total of all reporting groups
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID | Total
Number analyzed (Participants) | 126 | 252 | 253 | 631
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (18.11) | 36.8 (19.06) | 33.7 (17.15) | 35.2 (18.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 154 | 158 | 391
  Male | 47 | 98 | 95 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 30 | 37 | 88
  Not Hispanic or Latino | 104 | 218 | 212 | 534
  Unknown or Not Reported | 1 | 4 | 4 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 8 | 10 | 14 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 0 | 3
  Black or African American | 29 | 55 | 56 | 140
  White | 85 | 173 | 177 | 435
  Other | 4 | 9 | 6 | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms per square metre (kg/m^2)] | 26.92 (6.245) | 27.33 (6.745) | 27.47 (8.077) | 27.30 (7.212)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Investigator's Global Assessment - Treatment Success (IGA-TS) at Week 8
Description: The IGA is an overall eczema severity rating on a 5-point scale ranging from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, induration/papulation, and oozing/crusting. The IGA-TS is defined as an IGA score of 0 (clear skin) or 1 (almost clear skin) with ≥ 2 grade improvement from Baseline.
Time Frame: Baseline to Week 8
Population: ITT population included all participants who were randomized to the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants | 15.1 [9.3 to 22.5] | 50.0 [43.7 to 56.3] | 53.8 [47.4 to 60.0]
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Test type: Superiority; p < 0.0001, Exact Logistic Regression — The unadjusted p-values between each treatment group and vehicle were calculated based on Exact Logistic Regression including treatment and stratification factors to test the treatment difference; Odds Ratio (OR) = 6.38, 95% CI 2-sided [3.556 to 11.923]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Test type: Superiority; p < 0.0001, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.50, 95% CI 2-sided [4.178 to 14.040]

2. Secondary Outcome: VC Period: Percentage of Participants Who Achieved Eczema Area and Severity Index 75 (EASI75)
Description: EASI scoring system examines 4 areas of the body and weights them for participants of at least 8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l) for an average degree of severity of each sign in each region. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. An EASI75 responder was defined as a participant achieving 75% or greater improvement from Baseline in EASI score.
Time Frame: Baseline to Week 8
Population: ITT population included all participants who were randomized to the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants | 24.6 [17.4 to 33.1] | 56.0 [49.6 to 62.2] | 62.1 [55.8 to 68.1]
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Test type: Superiority; p < 0.0001, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.04, 95% CI 2-sided [2.441 to 6.808]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Test type: Superiority; p < 0.0001, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.22, 95% CI 2-sided [3.145 to 8.831]

3. Secondary Outcome: VC Period: Percentage of Participants With a ≥ 4-Point Improvement in Itch Numerical Rating Scale (NRS) Score
Description: The Itch NRS is a daily participant-reported measure (24-hour recall), using a diary, of the worst level of itch intensity. Participants were asked to rate the itching severity because of their AD in the daily diary by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best described their worst level of itching in the past 24 hours.
Time Frame: Baseline to Week 8
Population: ITT population included all participants who were randomized to the study. Number analyzed included participants in the ITT population with a Baseline Itch NRS score ≥ 4.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 78 | 156 | 161
percentage of participants | 15.4 | 40.4 | 52.2
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Test type: Superiority; p = 0.0002, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.66, 95% CI 2-sided [1.773 to 8.083]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Test type: Superiority; p < 0.0001, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.01, 95% CI 2-sided [2.931 to 13.220]

4. Secondary Outcome: VC Period: Percentage of Participants With a Clinically Meaningful (≥ 6-Point) Improvement in the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form - Sleep Disturbance (8b - 24-Hour Recall) Score
Description: The PROMIS Short Form - Sleep Disturbance (8b) questionnaire assesses participant's self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. It is a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep disturbance. Each item asks the participant to rate the severity of the participant's sleep disturbance.
Time Frame: Baseline to Week 8
Population: ITT population included all participants who were randomized to the study. Number analyzed included participants in the ITT population with a Baseline score ≥ 6.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 116 | 233 | 238
percentage of participants | 9.5 | 21.0 | 22.3
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Test type: Superiority; p = 0.0081, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.242 to 5.723]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0039, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.334 to 6.083]

5. Secondary Outcome: VC Period: Percentage of Participants With a Clinically Meaningful (≥ 6-Point) Improvement in the PROMIS Short Form - Sleep-Related Impairment (8a - 24-Hour Recall)
Description: The PROMIS Short Form - Sleep-Related Impairment (8a) questionnaire assesses participant's self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. The questionnaire has 8 simple questions with a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep-related impairment. Each item asks the participant to rate the severity of the participant's sleep impairment.
Time Frame: Baseline to Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 114 | 233 | 245
percentage of participants | 13.2 | 20.2 | 21.6
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Test type: Superiority; p = 0.1421, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.862 to 3.391]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0746, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.949 to 3.665]

6. Secondary Outcome: VC Period: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) and Treatment-Emergent Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or an important medical event may be considered serious when, based on appropriate medical judgment, the event may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above. A TEAE or treatment emergent SAE is any AE or SAE either reported for first time or worsening of a pre-existing event after first dose of study drug.
Time Frame: From first dose up to Week 8
Population: Safety population included all randomized participants who applied at least 1 application of ruxolitinib cream or vehicle cream.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  TEAE | 34.9 | 29.0 | 29.2
  Treatment Emergent SAE | 1.6 | 0.4 | 0.8

7. Secondary Outcome: LTS Period: Percentage of Participants With at Least One TEAE and Treatment Emergent SAE
Description: as for outcome 6
Time Frame: From first dose date in LTS Period (Week 8) until last follow-up visit (up to 52 weeks)
Population: LTS evaluable population included all participants who applied ruxolitinib 0.75% or 1.5% cream at least once during the LTS Period.
Measure: Number; unit: percentage of participants
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 48 | 47 | 222 | 225
percentage of participants
  TEAE | 47.9 | 48.9 | 54.5 | 53.3
  Treatment Emergent SAE | 6.3 | 2.1 | 2.3 | 1.3

8. Secondary Outcome: VC Period: Percentage of Participants Who Achieved an IGA-TS at Weeks 2 and 4
Description: The IGA is an overall eczema severity rating on a 0 (clear skin) to 4 (severe disease) scale. The score is based on an overall assessment of the degree of erythema, induration/papulation, and oozing/crusting. The IGA-TS is defined as an IGA score of 0 (clear skin) or 1 (almost clear skin) with ≥ 2 grade improvement from Baseline.
Time Frame: Baseline to Weeks 2 and 4
Population: ITT population included all participants who were randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  Week 2 | 3.2 | 22.2 | 27.3
  Week 4 | 6.3 | 42.5 | 46.6

9. Secondary Outcome: VC Period: Percentage of Participants Achieving IGA Scores of 0 or 1
Description: The IGA is an overall eczema severity rating on a 5-point scale ranging from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, induration/papulation, and oozing/crusting. IGA score signifies 0 (clear skin) and 1 (almost clear skin).
Time Frame: Weeks 2, 4 and 8
Population: ITT population included all participants who were randomized to the study.
Measure: Number; unit: percentage of participants
Groups:
- VC Period: Vehicle Cream BID: Participants received vehicle cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 8 during the VC Period.
- VC Period: Ruxolitinib 0.75% Cream BID: Participants received ruxolitinib 0.75% cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 8 during the VC Period.
- VC Period: Ruxolitinib 1.5% Cream BID: Participants received ruxolitinib 1.5% cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 8 during the VC Period.
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  Week 2 | 6.3 | 32.5 | 34.8
  Week 4 | 15.1 | 53.2 | 54.9
  Week 8 | 23.8 | 58.7 | 62.8

10. Secondary Outcome: LTS Period: Percentage of Participants Achieving IGA Scores of 0 or 1
Description: The IGA is an overall eczema severity rating on a 0 (clear skin) to 4 (severe disease) scale. The score is based on an overall assessment of the degree of erythema, induration/papulation, and oozing/crusting. IGA score signifies 0 (clear skin) and 1 (almost clear skin).
Time Frame: Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: LTS evaluable population included all participants who applied ruxolitinib 0.75% or 1.5% cream at least once during the LTS Period. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 48 | 47 | 222 | 225
percentage of participants
  Week 8 | 18.8 | 38.3 | 65.3 | 68.4
  Week 12: number analyzed (Participants) | 45 | 46 | 212 | 212
  Week 12 | 55.6 | 65.2 | 62.7 | 66.5
  Week 16: number analyzed (Participants) | 43 | 45 | 206 | 206
  Week 16 | 60.5 | 62.2 | 66.5 | 68.9
  Week 20: number analyzed (Participants) | 44 | 46 | 197 | 204
  Week 20 | 63.6 | 67.4 | 62.4 | 73.5
  Week 24: number analyzed (Participants) | 42 | 42 | 176 | 189
  Week 24 | 71.4 | 78.6 | 67.0 | 76.7
  Week 28: number analyzed (Participants) | 37 | 43 | 171 | 172
  Week 28 | 64.9 | 74.4 | 67.3 | 77.3
  Week 32: number analyzed (Participants) | 35 | 43 | 165 | 170
  Week 32 | 77.1 | 81.4 | 71.5 | 75.9
  Week 36: number analyzed (Participants) | 34 | 39 | 161 | 173
  Week 36 | 73.5 | 82.1 | 74.5 | 71.7
  Week 40: number analyzed (Participants) | 32 | 39 | 162 | 163
  Week 40 | 81.3 | 79.5 | 73.5 | 75.5
  Week 44: number analyzed (Participants) | 33 | 37 | 167 | 172
  Week 44 | 84.8 | 86.5 | 74.3 | 76.2
  Week 48: number analyzed (Participants) | 36 | 38 | 167 | 160
  Week 48 | 72.2 | 76.3 | 74.3 | 73.8
  Week 52: number analyzed (Participants) | 38 | 38 | 173 | 171
  Week 52 | 76.3 | 73.7 | 76.9 | 75.4

11. Secondary Outcome: VC Period: Percentage of Participants With a ≥ 4-Point Improvement in Itch NRS Score From Baseline to Weeks 2 and 4
Description: The Itch NRS is a daily participant-reported measure (24-hour recall), using a diary, of the worst level of itch intensity. Participants are asked to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes their worst level of itching in the past 24 hours.
Time Frame: Baseline to Weeks 2 and 4
Population: ITT population included all participants who were randomized to the study. Number analyzed includes participants in the ITT population with a Baseline Itch NRS score ≥ 4.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 78 | 156 | 161
percentage of participants
  Week 2 | 5.1 | 26.3 | 33.5
  Week 4 | 11.5 | 38.5 | 51.6

12. Secondary Outcome: VC Period: Percentage of Participants Achieving EASI50
Description: EASI scoring system examines 4 areas of the body and weights them for participants of at least 8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l) for an average degree of severity of each sign in each region. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. An EASI50 responder was defined as a participant achieving 50% or greater improvement from Baseline in EASI score.
Time Frame: Weeks 2, 4 and 8
Population: ITT population included all participants who were randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  Week 2 | 19.8 | 53.2 | 62.5
  Week 4 | 27.8 | 68.7 | 75.5
  Week 8 | 43.7 | 69.4 | 77.9

13. Secondary Outcome: VC Period: Percentage of Participants Achieving EASI75
Description: as for outcome 2
Time Frame: Weeks 2 and 4
Population: ITT population included all participants who were randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  Week 2 | 5.6 | 30.2 | 36.0
  Week 4 | 14.3 | 51.6 | 58.5

14. Secondary Outcome: VC Period: Percentage of Participants Achieving EASI90
Description: EASI scoring system examines 4 areas of the body and weights them for participants of at least 8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l) for an average degree of severity of each sign in each region. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. An EASI90 responder was defined as a participant achieving 90% or greater improvement from Baseline in EASI score.
Time Frame: Weeks 2, 4 and 8
Population: ITT population included all participants who were randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  Week 2 | 2.4 | 12.7 | 19.8
  Week 4 | 4.0 | 30.6 | 36.4
  Week 8 | 9.5 | 38.1 | 44.3

15. Secondary Outcome: VC Period: Percent Change From Baseline in EASI Score
Description: EASI scoring system examines 4 areas of the body and weights them for participants of at least 8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l) for an average degree of severity of each sign in each region. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4 and 8
Population: ITT population included all participants who were randomized to the study. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percent change
  Percent Change From Baseline at Week 2: number analyzed (Participants) | 115 | 239 | 242
  Percent Change From Baseline at Week 2 | -16.34 (3.42) | -51.82 (2.36) | -56.62 (2.35)
  Percent Change From Baseline at Week 4: number analyzed (Participants) | 108 | 237 | 242
  Percent Change From Baseline at Week 4 | -23.03 (3.90) | -68.04 (2.66) | -71.08 (2.64)
  Percent Change From Baseline at Week 8: number analyzed (Participants) | 101 | 225 | 232
  Percent Change From Baseline at Week 8 | -37.88 (3.72) | -71.01 (2.52) | -77.40 (2.49)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent change from Baseline in EASI score at Week 2; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -35.48, 95% CI 2-sided [-43.64 to -27.32], Standard Error of Mean 4.16
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent change from Baseline in EASI score at Week 2; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Method of Mean Difference] = -40.29, 95% CI 2-sided [-48.44 to -32.13], Standard Error of Mean 4.15
Statistical Analysis 3: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent change from Baseline in EASI score at Week 4; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -45.01, 95% CI 2-sided [-54.28 to -35.74], Standard Error of Mean 4.72
Statistical Analysis 4: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent change from Baseline in EASI score at Week 4; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -48.05, 95% CI 2-sided [-57.30 to -38.79], Standard Error of Mean 4.71
Statistical Analysis 5: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent change from Baseline in EASI score at Week 8; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures — The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -33.13, 95% CI 2-sided [-41.95 to -24.30], Standard Error of Mean 4.49
Statistical Analysis 6: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent change from Baseline in EASI score at Week 8; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -39.52, 95% CI 2-sided [-48.32 to -30.72], Standard Error of Mean 4.48

16. Secondary Outcome: VC Period: Percent Change From Baseline In SCORing Atopic Dermatitis (SCORAD) Score
Description: The SCORAD is a tool to assess extent and severity of eczema. To determine the extent, the rule of nines or handprint method is used to assess eczema affected area (A). To determine disease severity (B) it evaluates 6 clinical characteristics: 1. redness, 2. swelling, 3. oozing/crusting, 4. scratch marks, 5. lichenification, and 6. dryness on a 4-point scale of 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), added to give B with maximum score of 18. Subjective symptoms (C) of itch and sleeplessness are assessed using a visual analogue scale where 0 is no itch (or no sleeplessness) and 10 is the worst imaginable itch (or sleeplessness), added to give C with maximum score of 20. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combined using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4 and 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percent change
  Percent Change From Baseline at Week 2: number analyzed (Participants) | 115 | 239 | 242
  Percent Change From Baseline at Week 2 | -16.67 (34.152) | -43.96 (28.548) | -49.32 (31.878)
  Percent Change From Baseline at Week 4: number analyzed (Participants) | 107 | 237 | 241
  Percent Change From Baseline at Week 4 | -27.68 (34.518) | -57.80 (28.635) | -61.33 (30.113)
  Percent Change From Baseline at Week 8: number analyzed (Participants) | 101 | 225 | 230
  Percent Change From Baseline at Week 8 | -37.00 (36.392) | -62.14 (31.108) | -67.24 (28.711)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent change from Baseline in SCORAD score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; P-value was analyzed using ANCOVA model with treatment, stratification factors and Baseline score as covariates if applicable; Least Squares Mean Difference = -25.3, 95% CI 2-sided [-32.62 to -17.95], Standard Error of Mean 3.74
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent change from Baseline in SCORAD score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -30.4, 95% CI 2-sided [-37.68 to -23.06], Standard Error of Mean 3.72

17. Secondary Outcome: VC Period: Change From Baseline in Itch NRS Score
Description: The Itch NRS is a daily participant-reported measure (24-hour recall), using a diary, of the worst level of itch intensity. Participants are asked to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes their worst level of itching in the past 24 hours. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 98 | 210 | 220
  Change From Baseline at Week 2 | -0.89 (0.20) | -2.28 (0.14) | -2.53 (0.13)
  Change From Baseline at Week 4: number analyzed (Participants) | 94 | 214 | 219
  Change From Baseline at Week 4 | -1.08 (0.23) | -2.79 (0.16) | -3.16 (0.15)
  Change From Baseline at Week 8: number analyzed (Participants) | 80 | 185 | 203
  Change From Baseline at Week 8 | -1.54 (0.25) | -3.14 (0.17) | -3.53 (0.16)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in Itch NRS score at Week 2; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.39, 95% CI 2-sided [-1.87 to -0.91], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in Itch NRS score at Week 2; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.64, 95% CI 2-sided [-2.11 to -1.16], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in Itch NRS score at Week 4; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.70, 95% CI 2-sided [-2.25 to -1.15], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in Itch NRS score at Week 4; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -2.08, 95% CI 2-sided [-2.63 to -1.53], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in Itch NRS score at Week 8; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.60, 95% CI 2-sided [-2.20 to -1.01], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in Itch NRS score at Week 8; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.99, 95% CI 2-sided [-2.58 to -1.40], Standard Error of Mean 0.30

18. Secondary Outcome: VC Period: Time to Achieve Itch NRS Score Improvement of at Least 2, 3, or 4 Points
Description: The Itch NRS is a daily participant-reported measure (24-hour recall), using a diary, of the worst level of itch intensity. Participants were asked to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes their worst level of itching in the past 24 hours. Kaplan-Meier estimation method was used for analyses.
Time Frame: Up to Week 8
Population: ITT population included all participants who were randomized to the study. Number analyzed included participants in the ITT population with a Baseline Itch NRS score ≥ 2, ≥ 3 or ≥ 4 and a daily Itch NRS assessment during the VC Period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
days
  ≥ 2-Point Improvement in Itch NRS Score: number analyzed (Participants) | 105 | 212 | 220
  ≥ 2-Point Improvement in Itch NRS Score | 15.0 [10.0 to 22.0] | 4.0 [3.0 to 5.0] | 3.0 [3.0 to 4.0]
  ≥ 3-Point Improvement in Itch NRS Score: number analyzed (Participants) | 87 | 191 | 186
  ≥ 3-Point Improvement in Itch NRS Score | 27.0 [13.0 to 69.0] | 8.0 [7.0 to 11.0] | 6.0 [5.0 to 9.0]
  ≥ 4-Point Improvement in Itch NRS Score: number analyzed (Participants) | 78 | 156 | 161
  ≥ 4-Point Improvement in Itch NRS Score | NA [28.0 to NA] — The median time and upper limit of CI was not estimable due to low number of participants with data. | 14.0 [9.0 to 19.0] | 13.0 [9.0 to 15.0]

19. Secondary Outcome: VC Period: Change From Baseline in Skin Pain NRS Score
Description: The Skin Pain NRS is a daily patient-reported measure (24-hour recall), using a diary, of the worst level of pain intensity from 0 (no pain) to 10 (worst imaginable pain). Participants will be asked, "Rate the pain severity from your atopic dermatitis skin changes by selecting a number that best describes your worst level of pain in the past 24 hours." A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 97 | 210 | 219
  Change From Baseline at Week 2 | -0.70 (1.746) | -1.90 (1.950) | -2.07 (2.164)
  Change From Baseline at Week 4: number analyzed (Participants) | 94 | 213 | 219
  Change From Baseline at Week 4 | -0.84 (2.307) | -2.36 (2.217) | -2.72 (2.513)
  Change From Baseline at Week 8: number analyzed (Participants) | 80 | 185 | 201
  Change From Baseline at Week 8 | -1.16 (2.610) | -2.55 (2.360) | -2.84 (2.743)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in Skin Pain NRS score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-1.74 to -0.74], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in Skin Pain NRS score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -1.6, 95% CI 2-sided [-2.11 to -1.13], Standard Error of Mean 0.25

20. Secondary Outcome: VC Period: Percentage of Participants With a Clinically Meaningful (≥ 6-Point) Improvement in the PROMIS Short Form - Sleep Disturbance (8b) 24-Hour Recall Score
Description: The PROMIS Short Form - Sleep Disturbance (8b) questionnaire assesses participant's self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This questionnaire is completed in the morning by the participant where each item asks the participant to rate the severity of the participant's sleep disturbance. It is a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep disturbance.
Time Frame: Weeks 2 and 4
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 116 | 233 | 238
percentage of participants
  Week 2 | 5.2 | 13.7 | 14.7
  Week 4 | 6.9 | 19.3 | 21.0

21. Secondary Outcome: VC Period: Percentage of Participants With a Clinically Meaningful (≥ 6-Point) Improvement in the PROMIS Short Form - Sleep-Related Impairment (8a) 24-Hour Recall Score
Description: The PROMIS Short Form - Sleep-Related Impairment (8a) questionnaire assesses participant's self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. The questionnaire is filled in the evening where each item asks the participant to rate the severity of the participant's sleep impairment. It has 8 simple questions with a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep-related impairment.
Time Frame: Weeks 2 and 4
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 114 | 233 | 245
percentage of participants
  Week 2 | 8.8 | 16.3 | 13.5
  Week 4 | 13.2 | 20.6 | 19.2

22. Secondary Outcome: VC Period: Change From Baseline in PROMIS Short Form - Sleep Disturbance (8b) 24-Hour Recall Score
Description: The PROMIS Short Form - Sleep Disturbance (8b) questionnaire assesses participant's self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This questionnaire is completed in the morning by the participant where each item asks the participant to rate the severity of the participant's sleep disturbance. It is a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep disturbance. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 97 | 205 | 217
  Change From Baseline at Week 2 | -0.18 (0.45) | -1.72 (0.31) | -2.49 (0.30)
  Change From Baseline at Week 4: number analyzed (Participants) | 95 | 212 | 217
  Change From Baseline at Week 4 | -0.25 (0.50) | -2.58 (0.34) | -3.10 (0.33)
  Change From Baseline at Week 8: number analyzed (Participants) | 78 | 190 | 194
  Change From Baseline at Week 8 | -0.43 (0.59) | -2.97 (0.39) | -3.62 (0.39)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in PROMIS Short Form-Sleep Disturbance (8b) 24-hour recall score at Week 2; Test type: Superiority; p = 0.0049, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.53, 95% CI 2-sided [-2.60 to -0.47], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in PROMIS Short Form-Sleep Disturbance (8b) 24-hour recall score at Week 2; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -2.31, 95% CI 2-sided [-3.37 to -1.25], Standard Error of Mean 0.54
Statistical Analysis 3: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in PROMIS Short Form-Sleep Disturbance (8b) 24-hour recall score at Week 4; Test type: Superiority; p = 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -2.33, 95% CI 2-sided [-3.52 to -1.15], Standard Error of Mean 0.60
Statistical Analysis 4: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in PROMIS Short Form-Sleep Disturbance (8b) 24-hour recall score at Week 4; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -2.85, 95% CI 2-sided [-4.03 to -1.67], Standard Error of Mean 0.60
Statistical Analysis 5: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in PROMIS Short Form-Sleep Disturbance (8b) 24-hour recall score at Week 8; Test type: Superiority; p = 0.0004, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -2.54, 95% CI 2-sided [-3.93 to -1.14], Standard Error of Mean 0.71
Statistical Analysis 6: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in PROMIS Short Form-Sleep Disturbance (8b) 24-hour recall score at Week 8; Test type: Superiority; p < 0.0001, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -3.18, 95% CI 2-sided [-4.57 to -1.79], Standard Error of Mean 0.71

23. Secondary Outcome: VC Period: Change From Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-Hour Recall Score
Description: The PROMIS Short Form - Sleep-Related Impairment (8a) questionnaire assesses participant's self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. The questionnaire is filled in the evening where each item asks the participant to rate the severity of the participant's sleep impairment. It has 8 simple questions with a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep-related impairment. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 98 | 211 | 220
  Change From Baseline at Week 2 | -0.58 (0.49) | -1.76 (0.33) | -2.25 (0.33)
  Change From Baseline at Week 4: number analyzed (Participants) | 94 | 212 | 220
  Change From Baseline at Week 4 | -1.06 (0.55) | -2.71 (0.37) | -2.97 (0.36)
  Change From Baseline at Week 8: number analyzed (Participants) | 80 | 185 | 203
  Change From Baseline at Week 8 | -1.22 (0.62) | -3.34 (0.41) | -3.52 (0.40)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-hour recall score at Week 2; Test type: Superiority; p = 0.0487, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.18, 95% CI 2-sided [-2.35 to -0.01], Standard Error of Mean 0.60
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-hour recall score at Week 2; Test type: Superiority; p = 0.0049, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.68, 95% CI 2-sided [-2.84 to -0.51], Standard Error of Mean 0.59
Statistical Analysis 3: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-hour recall score at Week 4; Test type: Superiority; p = 0.0128, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.64, 95% CI 2-sided [-2.94 to -0.35], Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-hour recall score at Week 4; Test type: Superiority; p = 0.0037, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -1.91, 95% CI 2-sided [-3.20 to -0.62], Standard Error of Mean 0.66
Statistical Analysis 5: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-hour recall score at Week 8; Test type: Superiority; p = 0.0048, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -2.11, 95% CI 2-sided [-3.58 to -0.65], Standard Error of Mean 0.75
Statistical Analysis 6: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-hour recall score at Week 8; Test type: Superiority; p = 0.0020, Mixed-Model with Repeated Measures; The MMRM included the fixed effect of treatment, stratification factor, the visit, and treatment by visit interaction; Least Squares Mean Difference = -2.30, 95% CI 2-sided [-3.75 to -0.84], Standard Error of Mean 0.74

24. Secondary Outcome: LTS Period: Change From Baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 7-Day Recall Score
Description: as for outcome 23
Time Frame: Baseline, Weeks 12, 24, and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 48 | 47 | 222 | 225
score on a scale
  Change From Baseline at Week 12: number analyzed (Participants) | 41 | 45 | 198 | 198
  Change From Baseline at Week 12 | -1.51 (4.739) | -2.22 (7.305) | -0.39 (3.984) | -0.39 (3.907)
  Change From Baseline at Week 24: number analyzed (Participants) | 41 | 41 | 168 | 179
  Change From Baseline at Week 24 | -0.54 (5.211) | -2.66 (7.268) | 0.11 (4.929) | 0.02 (5.584)
  Change From Baseline at Week 52: number analyzed (Participants) | 37 | 36 | 168 | 167
  Change From Baseline at Week 52 | -0.97 (5.085) | -2.81 (7.005) | -0.37 (5.775) | -0.54 (5.511)

25. Secondary Outcome: LTS Period: Change From Baseline in PROMIS Short Form - Sleep Disturbance (8b) 7-Day Recall Score
Description: as for outcome 22
Time Frame: Baseline, Weeks 12, 24, and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 48 | 47 | 222 | 225
score on a scale
  Change From Baseline at Week 12: number analyzed (Participants) | 41 | 45 | 198 | 198
  Change From Baseline at Week 12 | -1.93 (5.284) | -2.67 (7.160) | -0.67 (4.575) | -0.66 (3.865)
  Change From Baseline at Week 24: number analyzed (Participants) | 41 | 41 | 168 | 179
  Change From Baseline at Week 24 | -1.22 (5.681) | -3.15 (8.242) | 0.02 (5.536) | 0.51 (5.563)
  Change From Baseline at Week 52: number analyzed (Participants) | 37 | 36 | 168 | 167
  Change From Baseline at Week 52 | -1.95 (4.876) | -3.31 (7.082) | -0.27 (6.506) | -0.07 (5.918)

26. Secondary Outcome: VC Period: Change From Baseline in Atopic Dermatitis Afflicted Percentage of Body Surface Area (%BSA)
Description: Body surface area affected by AD was assessed for 4 separate body regions and is collected as part of the EASI assessment: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region was assessed for disease extent ranging from 0% to 100% involvement. The overall total percentage was reported based off of all 4 body regions combined, after applying specific multipliers to the different body regions to account for the percent of the total BSA represented by each of the 4 regions. Used the percentage of skin affected for each region (0 to 100%) in EASI as follows: BSA Total = 0.1*BSA head and neck + 0.3*BSA trunk + 0.2* BSA upper limbs + 0.4*BSA lower limbs. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4 and 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
% BSA
  Change From Baseline at Week 2: number analyzed (Participants) | 115 | 239 | 242
  Change From Baseline at Week 2 | -0.43 (5.559) | -3.69 (4.230) | -3.76 (4.238)
  Change From Baseline at Week 4: number analyzed (Participants) | 108 | 237 | 242
  Change From Baseline at Week 4 | -1.56 (4.088) | -5.29 (4.969) | -5.25 (5.190)
  Change From Baseline at Week 8: number analyzed (Participants) | 101 | 225 | 232
  Change From Baseline at Week 8 | -2.51 (4.722) | -6.30 (5.378) | -6.54 (4.967)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in %BSA at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-4.07 to -2.18], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in %BSA at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -3.7, 95% CI 2-sided [-4.67 to -2.79], Standard Error of Mean 0.48

27. Secondary Outcome: LTS Period: Change From Baseline in Atopic Dermatitis Afflicted %BSA
Description: as for outcome 26
Time Frame: Baseline, Weeks 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 48 | 47 | 222 | 225
% BSA
  Change From Baseline at Week 12: number analyzed (Participants) | 44 | 46 | 212 | 212
  Change From Baseline at Week 12 | -4.23 (4.849) | -2.84 (4.907) | -6.84 (4.852) | -6.96 (4.989)
  Change From Baseline at Week 16: number analyzed (Participants) | 42 | 45 | 206 | 206
  Change From Baseline at Week 16 | -4.96 (5.194) | -2.98 (5.429) | -7.36 (4.875) | -7.26 (5.080)
  Change From Baseline at Week 20: number analyzed (Participants) | 44 | 46 | 197 | 204
  Change From Baseline at Week 20 | -4.78 (5.095) | -3.75 (5.321) | -7.69 (4.901) | -7.49 (5.012)
  Change From Baseline at Week 24: number analyzed (Participants) | 42 | 42 | 178 | 189
  Change From Baseline at Week 24 | -5.32 (4.964) | -3.85 (5.223) | -7.64 (4.998) | -7.64 (4.737)
  Change From Baseline at Week 28: number analyzed (Participants) | 37 | 43 | 171 | 172
  Change From Baseline at Week 28 | -4.56 (5.486) | -4.43 (4.995) | -7.66 (5.029) | -7.62 (4.913)
  Change From Baseline at Week 32: number analyzed (Participants) | 35 | 43 | 164 | 170
  Change From Baseline at Week 32 | -5.17 (4.472) | -4.53 (5.399) | -7.80 (5.011) | -7.61 (5.261)
  Change From Baseline at Week 36: number analyzed (Participants) | 34 | 39 | 161 | 173
  Change From Baseline at Week 36 | -5.21 (4.972) | -4.39 (5.509) | -8.18 (5.111) | -7.97 (5.010)
  Change From Baseline at Week 40: number analyzed (Participants) | 32 | 39 | 162 | 164
  Change From Baseline at Week 40 | -4.67 (5.519) | -4.75 (5.337) | -8.07 (4.899) | -8.11 (4.997)
  Change From Baseline at Week 44: number analyzed (Participants) | 33 | 37 | 168 | 172
  Change From Baseline at Week 44 | -5.28 (5.173) | -4.56 (5.609) | -8.14 (4.789) | -8.02 (4.939)
  Change From Baseline at Week 48: number analyzed (Participants) | 36 | 38 | 167 | 161
  Change From Baseline at Week 48 | -5.65 (5.128) | -4.58 (5.696) | -8.39 (5.023) | -7.96 (4.993)
  Change From Baseline at Week 52: number analyzed (Participants) | 38 | 38 | 173 | 171
  Change From Baseline at Week 52 | -5.72 (5.481) | -4.93 (5.771) | -8.58 (5.013) | -8.14 (4.906)

28. Secondary Outcome: VC Period: Change From Baseline in Patient-Oriented Eczema Measure (POEM) Score
Description: The POEM is a 7-question quality-of-life assessment that asks how many days the participant has been bothered by various aspects of their skin condition during the past 7 days. It assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (clear or almost clear) to 28 (very severe eczema). High scores are indicative of more severe disease and poor quality of life. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 112 | 236 | 237
  Change From Baseline at Week 2 | -2.25 (5.779) | -9.47 (7.212) | -10.60 (6.670)
  Change From Baseline at Week 4: number analyzed (Participants) | 106 | 234 | 240
  Change From Baseline at Week 4 | -3.38 (6.685) | -10.12 (7.380) | -11.53 (6.891)
  Change From Baseline at Week 8: number analyzed (Participants) | 99 | 222 | 228
  Change From Baseline at Week 8 | -4.30 (7.044) | -10.60 (7.262) | -11.82 (6.931)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in POEM score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -5.1, 95% CI 2-sided [-6.43 to -3.80], Standard Error of Mean 0.67
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in POEM score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -6.3, 95% CI 2-sided [-7.62 to -5.00], Standard Error of Mean 0.67

29. Secondary Outcome: LTS Period: Change From Baseline in POEM Score
Description: The POEM is a 7-question quality-of-life assessment that asks how many days the participant has been bothered by various aspects of their skin condition during the past 7 days. It assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 12, 24, and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 48 | 47 | 222 | 225
score on a scale
  Change From Baseline at Week 12: number analyzed (Participants) | 41 | 46 | 206 | 206
  Change From Baseline at Week 12 | -5.95 (6.607) | -6.89 (9.730) | -10.74 (6.653) | -11.38 (6.710)
  Change From Baseline at Week 24: number analyzed (Participants) | 41 | 42 | 173 | 185
  Change From Baseline at Week 24 | -4.46 (6.185) | -7.26 (9.189) | -10.46 (6.655) | -11.44 (6.689)
  Change From Baseline at Week 52: number analyzed (Participants) | 38 | 38 | 174 | 170
  Change From Baseline at Week 52 | -4.61 (6.868) | -7.00 (8.752) | -10.51 (7.396) | -10.61 (7.057)

30. Secondary Outcome: VC Period: Change From Baseline in Dermatology Life Quality Index (DLQI) Score
Description: The DLQI is a simple, 10 question (Q) validated quality-of-life questionnaire to measure how much the skin problem has affected the participant. It covers 6 domains including symptoms and feelings (Q1 and Q2), daily activities (Q3 and Q4), leisure (Q5 and Q6), work and school (Q7), personal relationships (Q8 and Q9), and treatment(Q10). The recall Period of this scale is over the last week. Response categories include 0-not at all, 1-a little, 2-a lot, and 3-very much, and unanswered or not relevant responses scored as 0. Scores range from 0 ("no impact on participant's life") to 30 ("extremely large effect on participant's life"), and a 4-point change from Baseline is considered as the minimal clinically important difference threshold. A negative change from Baseline indicates less impact of the skin problem on participant's life.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: ITT population included all participants who were randomized to the study. Participants in the ITT population with age >= 16 were included. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 107 | 215 | 223
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 94 | 200 | 209
  Change From Baseline at Week 2 | -1.54 (4.618) | -6.18 (5.740) | -6.90 (5.980)
  Change From Baseline at Week 4: number analyzed (Participants) | 88 | 198 | 211
  Change From Baseline at Week 4 | -2.50 (6.101) | -6.88 (5.867) | -7.15 (6.565)
  Change From Baseline at Week 8: number analyzed (Participants) | 82 | 188 | 201
  Change From Baseline at Week 8 | -2.83 (6.722) | -7.28 (5.907) | -7.72 (6.152)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in total DLQI score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -3.8, 95% CI 2-sided [-4.85 to -2.68], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in total DLQI score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -4.5, 95% CI 2-sided [-5.56 to -3.42], Standard Error of Mean 0.55

31. Secondary Outcome: LTS Period: Change From Baseline in DLQI Score
Description: as for outcome 30
Time Frame: Baseline, Weeks 12, 24, and 52
Population: LTS evaluable population included all participants who applied ruxolitinib 0.75% or 1.5% cream at least once during the LTS Period. Participants in the LTS evaluable population with age >= 16 were included. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 40 | 38 | 189 | 200
score on a scale
  Change From Baseline at Week 12: number analyzed (Participants) | 34 | 38 | 175 | 185
  Change From Baseline at Week 12 | -3.65 (5.602) | -4.53 (6.246) | -7.67 (5.855) | -7.79 (6.240)
  Change From Baseline at Week 24: number analyzed (Participants) | 33 | 34 | 148 | 167
  Change From Baseline at Week 24 | -3.21 (4.814) | -5.32 (6.304) | -7.87 (6.080) | -7.75 (6.277)
  Change From Baseline at Week 52: number analyzed (Participants) | 31 | 31 | 151 | 149
  Change From Baseline at Week 52 | -3.35 (5.438) | -4.81 (6.720) | -7.95 (6.589) | -7.70 (6.443)

32. Secondary Outcome: VC Period: Change From Baseline in Children Dermatology Life Quality Index (CDLQI) Score
Description: CDLQI is the youth/children's version of the DLQI. The CDLQI is a simple 10 question (Q) validated quality-of-life questionnaire. It covers 6 domains including symptoms and feelings (Q1 and Q2), leisure (Q4, Q5, and Q6), school or holidays (Q7), personal relationships (Q3 and Q8), sleep (Q9) and treatment (Q10). Response categories include 0-not at all, 1-a little, 2-a lot, and 3-very much, and unanswered or not relevant responses scored as 0. The total DLQI score is calculated by adding the score of each question resulting in a maximum score of 30 (extremely large effect on participant's life) and a minimum score of 0 (no impact on participant's life) and a 4-point change from Baseline is considered as the minimal clinically important difference threshold. A negative change from Baseline indicates less impact of the skin problem on participant's life.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: ITT population included all participants who were randomized to the study. Participants in the ITT population with age < 16 were included. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 19 | 37 | 30
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 18 | 33 | 29
  Change From Baseline at Week 2 | -1.06 (3.733) | -5.06 (6.937) | -6.76 (6.306)
  Change From Baseline at Week 4: number analyzed (Participants) | 17 | 34 | 29
  Change From Baseline at Week 4 | -2.47 (6.530) | -4.35 (8.683) | -6.90 (5.101)
  Change From Baseline at Week 8: number analyzed (Participants) | 16 | 33 | 28
  Change From Baseline at Week 8 | -2.31 (5.618) | -5.88 (7.524) | -7.61 (6.142)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in total CDLQI score at Week 8; Test type: Superiority; p = 0.0018, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -3.3, 95% CI 2-sided [-5.29 to -1.26], Standard Error of Mean 1.01
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in total CDLQI score at Week 8; Test type: Superiority; p = 0.0378, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -2.3, 95% CI 2-sided [-4.43 to -0.13], Standard Error of Mean 1.08

33. Secondary Outcome: LTS Period: Change From Baseline in CDLQI Score
Description: as for outcome 32
Time Frame: Baseline, Weeks 12, 24, and 52
Population: LTS evaluable population included all participants who applied ruxolitinib 0.75% or 1.5% cream at least once during the LTS Period. Participants in the LTS evaluable population with age < 16 were included. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 8 | 9 | 33 | 25
score on a scale
  Change From Baseline at Week 12: number analyzed (Participants) | 6 | 8 | 30 | 22
  Change From Baseline at Week 12 | -4.00 (5.477) | -1.13 (8.097) | -5.83 (7.661) | -8.86 (5.532)
  Change From Baseline at Week 24: number analyzed (Participants) | 7 | 8 | 25 | 19
  Change From Baseline at Week 24 | -2.71 (5.155) | -2.00 (3.780) | -6.72 (7.640) | -9.42 (7.214)
  Change From Baseline at Week 52: number analyzed (Participants) | 6 | 7 | 23 | 21
  Change From Baseline at Week 52 | -4.33 (8.359) | -0.43 (4.928) | -6.70 (7.766) | -9.71 (6.262)

34. Secondary Outcome: VC Period: Mean Patient Global Impression of Change (PGIC) Score at Weeks 2, 4, and 8
Description: The PGIC is a participants' self-reporting measure that reflects their belief about the efficacy of treatment. It is a 7-point scale where participants rate the questions as: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The lower score indicates improvement.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Week 2: number analyzed (Participants) | 113 | 236 | 237
  Week 2 | 3.53 (1.500) | 2.06 (0.937) | 1.94 (0.911)
  Week 4: number analyzed (Participants) | 105 | 237 | 240
  Week 4 | 3.30 (1.434) | 1.78 (0.903) | 1.68 (0.843)
  Week 8: number analyzed (Participants) | 100 | 223 | 229
  Week 8 | 3.08 (1.489) | 1.76 (0.913) | 1.61 (0.914)

35. Secondary Outcome: VC Period: Percentage of Participants With Each Score on the PGIC at Weeks 2, 4, and 8
Description: as for outcome 34
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  Week 2 - Very Much Improved: 1: number analyzed (Participants) | 113 | 236 | 237
  Week 2 - Very Much Improved: 1 | 5.3 | 31.4 | 36.7
  Week 2 - Much Improved: 2: number analyzed (Participants) | 113 | 236 | 237
  Week 2 - Much Improved: 2 | 18.6 | 38.6 | 40.1
  Week 2 - Minimally Improved: 3: number analyzed (Participants) | 113 | 236 | 237
  Week 2 - Minimally Improved: 3 | 37.2 | 25.0 | 16.9
  Week 2 - No Change: 4: number analyzed (Participants) | 113 | 236 | 237
  Week 2 - No Change: 4 | 13.3 | 4.2 | 5.5
  Week 2 - Minimally Worse: 5: number analyzed (Participants) | 113 | 236 | 237
  Week 2 - Minimally Worse: 5 | 11.5 | 0.4 | 0.8
  Week 2 - Much Worse: 6: number analyzed (Participants) | 113 | 236 | 237
  Week 2 - Much Worse: 6 | 10.6 | 0.0 | 0.0
  Week 2 - Very Much Worse: 7: number analyzed (Participants) | 113 | 236 | 237
  Week 2 - Very Much Worse: 7 | 3.5 | 0.4 | 0.0
  Week 4 - Very Much Improved: 1: number analyzed (Participants) | 105 | 237 | 240
  Week 4 - Very Much Improved: 1 | 6.7 | 48.5 | 51.7
  Week 4 - Much Improved: 2: number analyzed (Participants) | 105 | 237 | 240
  Week 4 - Much Improved: 2 | 22.9 | 29.5 | 32.1
  Week 4 - Minimally Improved: 3: number analyzed (Participants) | 105 | 237 | 240
  Week 4 - Minimally Improved: 3 | 38.1 | 18.1 | 13.3
  Week 4 - No Change: 4: number analyzed (Participants) | 105 | 237 | 240
  Week 4 - No Change: 4 | 11.4 | 3.0 | 2.1
  Week 4 - Minimally Worse: 5: number analyzed (Participants) | 105 | 237 | 240
  Week 4 - Minimally Worse: 5 | 11.4 | 0.8 | 0.8
  Week 4 - Much Worse: 6: number analyzed (Participants) | 105 | 237 | 240
  Week 4 - Much Worse: 6 | 6.7 | 0.0 | 0.0
  Week 4 - Very Much Worse: 7: number analyzed (Participants) | 105 | 237 | 240
  Week 4 - Very Much Worse: 7 | 2.9 | 0.0 | 0.0
  Week 8 - Very Much Improved: 1: number analyzed (Participants) | 100 | 223 | 229
  Week 8 - Very Much Improved: 1 | 11.0 | 48.4 | 59.8
  Week 8 - Much Improved: 2: number analyzed (Participants) | 100 | 223 | 229
  Week 8 - Much Improved: 2 | 30.0 | 33.2 | 25.8
  Week 8 - Minimally Improved: 3: number analyzed (Participants) | 100 | 223 | 229
  Week 8 - Minimally Improved: 3 | 29.0 | 14.8 | 10.0
  Week 8 - No Change: 4: number analyzed (Participants) | 100 | 223 | 229
  Week 8 - No Change: 4 | 12.0 | 1.3 | 2.2
  Week 8 - Minimally Worse: 5: number analyzed (Participants) | 100 | 223 | 229
  Week 8 - Minimally Worse: 5 | 7.0 | 2.2 | 2.2
  Week 8 - Much Worse: 6: number analyzed (Participants) | 100 | 223 | 229
  Week 8 - Much Worse: 6 | 10.0 | 0.0 | 0.0
  Week 8 - Very Much Worse: 7: number analyzed (Participants) | 100 | 223 | 229
  Week 8 - Very Much Worse: 7 | 1.0 | 0.0 | 0.0

36. Secondary Outcome: VC Period: Percentage of Participants With a Score of Either 1 or 2 on the PGIC at Weeks 2, 4, and 8
Description: as for outcome 34
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
percentage of participants
  Week 2: number analyzed (Participants) | 113 | 236 | 237
  Week 2 | 23.9 [16.4 to 32.8] | 69.9 [63.6 to 75.7] | 76.8 [70.9 to 82.0]
  Week 4: number analyzed (Participants) | 105 | 237 | 240
  Week 4 | 29.5 [21.0 to 39.2] | 78.1 [72.2 to 83.2] | 83.8 [78.5 to 88.2]
  Week 8: number analyzed (Participants) | 100 | 223 | 229
  Week 8 | 41.0 [31.3 to 51.3] | 81.6 [75.9 to 86.5] | 85.6 [80.4 to 89.9]
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percentage of participants with a score of either 1 or 2 on the PGIC at Week 8; Test type: Superiority; p < 0.0001, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.28, 95% CI 2-sided [3.632 to 11.018]
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percentage of participants with a score of either 1 or 2 on the PGIC at Week 8; Test type: Superiority; p < 0.0001, Exact Logistic Regression — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 8.39, 95% CI 2-sided [4.755 to 15.083]

37. Secondary Outcome: VC Period: Change From Baseline in EuroQuality of Life Five Dimensions (EQ-5D-5L) Visual Analogue Scale (VAS) Score
Description: EQ-5D-5L questionnaire has 2 parts: EQ-5D-5L descriptive system & EQ-VAS. EQ-5D is a validated, self-administered, generic utility questionnaire wherein participants rate their current health state based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. 5L indicates that for each dimension, there are 5 levels:1=no problems,2=slight problems,3=moderate problems,4=severe problems, and 5=extreme problems. EQ-5D-5L score is assessed using VAS that ranges from 0 to 100 millimetres (mm), where 0 indicates "worst health you can imagine" and 100 indicates "best health you can imagine". The participant was asked to indicate his/her health state over past 7 days in each of the 5 dimensions. Digits for the 5 dimensions can be combined into a 5-digit number that describes the participant's health state. In the EQ-VAS, participants had to record their health state on a scale ranging from 0 to 100. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Change From Baseline at Week 2: number analyzed (Participants) | 114 | 237 | 237
  Change From Baseline at Week 2 | -0.94 (14.046) | 6.93 (17.690) | 8.21 (15.770)
  Change From Baseline at Week 4: number analyzed (Participants) | 107 | 237 | 241
  Change From Baseline at Week 4 | 1.76 (11.618) | 8.73 (17.494) | 7.10 (16.697)
  Change From Baseline at Week 8: number analyzed (Participants) | 100 | 223 | 229
  Change From Baseline at Week 8 | 1.74 (14.376) | 9.12 (17.871) | 7.98 (16.813)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Change from Baseline in EQ VAS score at Week 8; Test type: Superiority; p = 0.0037, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = 4.9, 95% CI 2-sided [1.59 to 8.15], Standard Error of Mean 1.67
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Change from Baseline in EQ VAS score at Week 8; Test type: Superiority; p = 0.0006, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = 5.7, 95% CI 2-sided [2.45 to 8.96], Standard Error of Mean 1.66

38. Secondary Outcome: VC Period: Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP) Version 2.0 (v2.0)
Description: The WPAI-SHP is a 6-item participant questionnaire developed to measure the effect of overall health and specific symptoms on productivity at work and regular activities outside of it in the past 7 days. The WPAI-SHP consists of 6 questions as follows: 1=currently employed; 2=hours missed due to AD; 3=hours missed other reasons; 4=hours actually worked; 5=degree AD affected productivity while working; 6=degree AD affected regular activities and the computed percentage, range for each sub scale is from 0 to 100, with higher values indicating greater impairment and less productivity. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC Period: Vehicle Cream BID | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 126 | 252 | 253
score on a scale
  Percent Work Time Missed Due to AD: Change From Baseline at Week 2: number analyzed (Participants) | 54 | 111 | 121
  Percent Work Time Missed Due to AD: Change From Baseline at Week 2 | 4.45 (19.542) | -3.89 (24.223) | 1.19 (14.954)
  Percent Work Time Missed Due to AD: Change From Baseline at Week 4: number analyzed (Participants) | 48 | 107 | 124
  Percent Work Time Missed Due to AD: Change From Baseline at Week 4 | 14.09 (30.660) | 1.22 (23.898) | 3.43 (17.242)
  Percent Work Time Missed Due to AD: Change From Baseline at Week 8: number analyzed (Participants) | 48 | 108 | 119
  Percent Work Time Missed Due to AD: Change From Baseline at Week 8 | 5.07 (23.253) | -0.26 (23.891) | 6.23 (22.211)
  Percent Impairment While Working Due to AD: Change From Baseline at Week 2: number analyzed (Participants) | 53 | 110 | 120
  Percent Impairment While Working Due to AD: Change From Baseline at Week 2 | -7.36 (22.630) | -15.00 (22.494) | -16.75 (20.951)
  Percent Impairment While Working Due to AD: Change From Baseline at Week 4: number analyzed (Participants) | 45 | 105 | 123
  Percent Impairment While Working Due to AD: Change From Baseline at Week 4 | -9.56 (25.580) | -16.86 (22.417) | -19.43 (20.933)
  Percent Impairment While Working Due to AD: Change From Baseline at Week 8: number analyzed (Participants) | 48 | 105 | 118
  Percent Impairment While Working Due to AD: Change From Baseline at Week 8 | -13.54 (28.019) | -19.43 (24.878) | -21.61 (22.071)
  Percent Overall Work Impairment Due to AD: Change From Baseline at Week 2: number analyzed (Participants) | 53 | 110 | 120
  Percent Overall Work Impairment Due to AD: Change From Baseline at Week 2 | -5.27 (21.539) | -15.04 (27.812) | -15.49 (23.785)
  Percent Overall Work Impairment Due to AD: Change From Baseline at Week 4: number analyzed (Participants) | 45 | 105 | 123
  Percent Overall Work Impairment Due to AD: Change From Baseline at Week 4 | -2.35 (27.602) | -13.82 (26.207) | -15.82 (25.545)
  Percent Overall Work Impairment Due to AD: Change From Baseline at Week 8: number analyzed (Participants) | 48 | 105 | 118
  Percent Overall Work Impairment Due to AD: Change From Baseline at Week 8 | -9.01 (31.735) | -18.09 (27.718) | -15.54 (27.119)
  Percent Activity Impairment Due to AD: Change From Baseline at Week 2: number analyzed (Participants) | 114 | 237 | 237
  Percent Activity Impairment Due to AD: Change From Baseline at Week 2 | -6.32 (23.434) | -16.58 (24.696) | -21.56 (24.695)
  Percent Activity Impairment Due to AD: Change From Baseline at Week 4: number analyzed (Participants) | 106 | 237 | 241
  Percent Activity Impairment Due to AD: Change From Baseline at Week 4 | -10.09 (26.349) | -20.80 (24.107) | -23.53 (25.422)
  Percent Activity Impairment Due to AD: Change From Baseline at Week 8: number analyzed (Participants) | 100 | 223 | 229
  Percent Activity Impairment Due to AD: Change From Baseline at Week 8 | -11.70 (28.992) | -21.30 (24.653) | -24.06 (26.682)
Statistical Analysis 1: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent work time missed due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p = 0.1417, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -4.9, 95% CI 2-sided [-11.49 to 1.65], Standard Error of Mean 3.34
Statistical Analysis 2: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent work time missed due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p = 0.6037, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -1.7, 95% CI 2-sided [-8.19 to 4.77], Standard Error of Mean 3.29
Statistical Analysis 3: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent impairment while working due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p = 0.0003, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -11.0, 95% CI 2-sided [-16.89 to -5.12], Standard Error of Mean 2.99
Statistical Analysis 4: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent impairment while working due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -12.2, 95% CI 2-sided [-17.98 to -6.47], Standard Error of Mean 2.93
Statistical Analysis 5: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent overall work impairment due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -15.4, 95% CI 2-sided [-22.95 to -7.81], Standard Error of Mean 3.85
Statistical Analysis 6: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent overall work impairment due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p = 0.0011, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -12.4, 95% CI 2-sided [-19.85 to -5.01], Standard Error of Mean 3.77
Statistical Analysis 7: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 0.75% Cream BID; Percent activity impairment due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -10.5, 95% CI 2-sided [-14.64 to -6.29], Standard Error of Mean 2.13
Statistical Analysis 8: Comparison: VC Period: Vehicle Cream BID vs VC Period: Ruxolitinib 1.5% Cream BID; Percent activity impairment due to AD: Change from Baseline in WPAI-SHP v2.0 at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; Least Squares Mean Difference = -12.4, 95% CI 2-sided [-16.60 to -8.29], Standard Error of Mean 2.12

39. Secondary Outcome: LTS Period: Change From Baseline in WPAI-SHP v2.0
Description: as for outcome 38
Time Frame: Baseline, Weeks 12, 24, 36, and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 48 | 47 | 222 | 225
score on a scale
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12: number analyzed (Participants) | 20 | 22 | 98 | 110
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12 | -4.78 (18.023) | -2.02 (4.902) | -0.26 (27.118) | 7.72 (22.067)
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24: number analyzed (Participants) | 19 | 18 | 78 | 94
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24 | -0.39 (21.466) | 4.77 (16.899) | -1.00 (28.511) | 4.96 (18.942)
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36: number analyzed (Participants) | 16 | 13 | 75 | 81
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36 | -3.92 (23.687) | -3.12 (6.143) | -0.32 (27.115) | 8.93 (21.916)
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52: number analyzed (Participants) | 13 | 12 | 81 | 82
  Percent Work Time Missed Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52 | -8.11 (18.718) | 3.23 (26.008) | 1.81 (26.094) | 2.38 (16.245)
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12: number analyzed (Participants) | 20 | 22 | 95 | 108
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12 | -11.50 (23.458) | -18.64 (28.668) | -20.21 (24.925) | -20.65 (21.844)
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24: number analyzed (Participants) | 19 | 18 | 77 | 93
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24 | -8.42 (16.754) | -16.67 (28.697) | -23.51 (25.067) | -23.66 (24.396)
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36: number analyzed (Participants) | 16 | 13 | 73 | 81
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36 | -3.13 (20.887) | -8.46 (33.378) | -23.15 (25.813) | -22.72 (23.185)
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52: number analyzed (Participants) | 13 | 12 | 79 | 83
  Percent Impairment While Working Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52 | -10.00 (25.166) | -20.00 (27.634) | -23.42 (26.597) | -22.77 (24.109)
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12: number analyzed (Participants) | 20 | 22 | 95 | 108
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12 | -12.18 (24.763) | -19.64 (28.842) | -18.21 (28.345) | -14.99 (28.777)
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24: number analyzed (Participants) | 19 | 18 | 76 | 93
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24 | -7.46 (16.254) | -12.96 (34.336) | -20.26 (31.191) | -18.60 (28.284)
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36: number analyzed (Participants) | 16 | 13 | 73 | 80
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36 | -5.70 (23.040) | -10.43 (33.034) | -20.52 (31.307) | -14.86 (29.482)
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52: number analyzed (Participants) | 13 | 12 | 79 | 82
  Percent Overall Work Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52 | -16.36 (29.721) | -16.67 (40.350) | -19.42 (29.878) | -20.50 (26.949)
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12: number analyzed (Participants) | 41 | 46 | 206 | 206
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 12 | -12.20 (21.273) | -8.48 (26.244) | -21.50 (26.470) | -25.19 (26.314)
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24: number analyzed (Participants) | 41 | 42 | 173 | 186
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 24 | -11.46 (16.517) | -7.14 (25.113) | -22.83 (27.440) | -27.47 (25.943)
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36: number analyzed (Participants) | 36 | 40 | 163 | 177
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 36 | -6.39 (18.997) | -1.25 (27.845) | -24.48 (26.203) | -26.84 (27.493)
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52: number analyzed (Participants) | 38 | 38 | 175 | 172
  Percent Activity Impairment Due to AD: Change From Baseline in WPAI-SHP v2.0 at Week 52 | -11.05 (24.910) | -13.42 (25.392) | -22.91 (27.669) | -26.92 (28.042)

40. Secondary Outcome: VC Period: Trough Plasma Concentrations of Ruxolitinib
Description: Plasma samples were collected just before the morning application of study drug during each specified time point.
Time Frame: Pre-dose at Weeks 2, 4 and 8
Population: The pharmacokinetic (PK) evaluable population included all participants who applied at least 1 application of ruxolitinib cream and provided at least 1 postdose plasma sample (1 PK measurement) that complies with the instruction in the Protocol. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: nanomole per liter (nM)
Arm/Group | VC Period: Ruxolitinib 0.75% Cream BID | VC Period: Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 236 | 241
nanomole per liter (nM)
  Week 2: number analyzed (Participants) | 227 | 230
  Week 2 | 26.8 (51.2) | 33.4 (49.9)
  Week 4: number analyzed (Participants) | 229 | 232
  Week 4 | 25.1 (42.7) | 34.7 (43.3)
  Week 8: number analyzed (Participants) | 218 | 224
  Week 8 | 24.0 (39.7) | 33.3 (49.5)

41. Secondary Outcome: LTS Period: Trough Plasma Concentrations of Ruxolitinib
Description: Plasma samples were collected just before the morning application of study drug during each specified time point.
Time Frame: Pre-dose at Weeks 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: The PK evaluable population included all participants who applied at least 1 application of ruxolitinib cream and provided at least 1 postdose plasma sample (1 PK measurement) that complies with the instruction in the Protocol. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | LTS Period: Vehicle Cream to Ruxolitinib 0.75% Cream BID | LTS Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID | LTS Period: Ruxolitinib 0.75% Cream | LTS Period: Ruxolitinib 1.5% Cream
Number analyzed (Participants) | 44 | 47 | 210 | 213
nM
  Week 12: number analyzed (Participants) | 42 | 45 | 208 | 207
  Week 12 | 13.8 (21.3) | 21.9 (34.4) | 16.5 (28.1) | 24.9 (45.4)
  Week 16: number analyzed (Participants) | 42 | 44 | 200 | 201
  Week 16 | 11.9 (18.8) | 18.1 (34.6) | 19.7 (58.8) | 24.6 (51.0)
  Week 20: number analyzed (Participants) | 43 | 46 | 193 | 199
  Week 20 | 13.0 (22.2) | 15.4 (32.0) | 16.1 (31.2) | 24.2 (46.1)
  Week 24: number analyzed (Participants) | 40 | 42 | 171 | 182
  Week 24 | 13.0 (22.1) | 18.7 (31.6) | 18.8 (42.4) | 24.6 (51.8)
  Week 28: number analyzed (Participants) | 34 | 43 | 164 | 170
  Week 28 | 18.5 (36.9) | 15.5 (24.6) | 16.2 (31.2) | 23.7 (45.3)
  Week 32: number analyzed (Participants) | 32 | 42 | 162 | 164
  Week 32 | 17.8 (27.3) | 17.7 (33.3) | 21.4 (59.8) | 21.0 (35.3)
  Week 36: number analyzed (Participants) | 33 | 38 | 155 | 169
  Week 36 | 21.1 (54.8) | 29.5 (84.0) | 15.7 (30.5) | 26.6 (51.2)
  Week 40: number analyzed (Participants) | 32 | 38 | 158 | 161
  Week 40 | 14.9 (25.3) | 16.5 (31.0) | 14.7 (27.6) | 23.2 (64.1)
  Week 44: number analyzed (Participants) | 32 | 37 | 160 | 168
  Week 44 | 14.3 (23.7) | 15.7 (32.6) | 17.3 (33.5) | 26.8 (58.6)
  Week 48: number analyzed (Participants) | 34 | 37 | 159 | 156
  Week 48 | 15.6 (26.8) | 17.9 (56.0) | 15.3 (30.3) | 24.8 (55.3)
  Week 52: number analyzed (Participants) | 36 | 38 | 167 | 166
  Week 52 | 11.0 (17.9) | 14.2 (27.5) | 11.9 (20.5) | 21.0 (55.7)

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Description: For safety analysis, participants who crossed over treatment from vehicle to active arm (0.75% BID and 1.5% BID Ruxolitinib cream) in LTS Period are counted both in vehicle arm and active arms in the number of participants summaries.
Groups:
- Vehicle Cream BID: Participants received vehicle cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 52 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
- Ruxolitinib 0.75% Cream BID: Participants received ruxolitinib 0.75% cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 52 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
- Ruxolitinib 1.5% Cream BID: Participants received ruxolitinib 1.5% cream, applied topically to the affected areas as a thin film BID from Day 1 to Week 52 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
Arm/Group | Vehicle Cream BID | Ruxolitinib 0.75% Cream BID | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 2/126 | 9/300 | 6/300
Other Adverse Events (participants affected / at risk) | 10/126 | 52/300 | 70/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Cream BID (N=126) | Ruxolitinib 0.75% Cream BID (N=300) | Ruxolitinib 1.5% Cream BID (N=300)
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Serositis (General disorders) | 0 | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Cream BID (N=126) | Ruxolitinib 0.75% Cream BID (N=300) | Ruxolitinib 1.5% Cream BID (N=300)
Nasopharyngitis (Infections and infestations) | 2 | 18 | 31
Upper respiratory tract infection (Infections and infestations) | 4 | 27 | 36
Headache (Nervous system disorders) | 5 | 11 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT03745638/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT03745638/SAP_001.pdf